CLINICAL TRIAL: NCT07219355
Title: Expanding Provider Capacity to Prevent Rural Veteran Suicide: Virtual Reality Lethal Means Safety Training
Brief Title: Virtual Reality Lethal Means Safety Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-0085; ECR-0-140-23 (Other Grant/Funding Number: American Foundation for Suicide Prevention)
Record Dates: First submitted 2025-09-23; First posted 2025-10-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Suicide, Attempted; Suicide, Completed; Suicide Prevention; Mental Health Training; Rural Health; Veterans
Keywords: Veterans; Rural Veterans; Suicide Prevention; Suicide Risk; Firearm Safety; Medication Safety; Lethal Means Safety Counseling; Virtual Reality (VR); VR Training Simulation; Rural Health
MeSH Terms: conditions — Suicide, Attempted; Suicide, Completed; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group behavioral clinical trial with two arms. Healthcare providers (≥18, serving Veterans in Texas) are prospectively assigned in a 1:1 ratio to:
  Intervention (VR-LMST): Participants use a Meta Quest 3 headset to complete an interactive virtual reality simulation of a rural clinic visit with a Veteran avatar at risk for suicide, practicing lethal means safety counseling (firearm and medication storage).
  Control (2D Video): Participants use the headset to view a 2D, ~10-minute video of the lethal means safety counseling training.
  Randomization is computer-generated (Excel) with no crossover. Masking is None (Open Label); outcome assessment uses standardized self-report instruments. Surveys are administered pre-intervention, post-intervention, and at 3-month follow-up (e.g., CALM Scale for confidence/comfortability/intentions; ITC-SOPI for presence/engagement/ecological validity/negative effects.
Masking Description: Participants and study personnel are aware of assignment because the intervention content differs (interactive VR simulation vs. 2D video). Both groups use headsets to reduce expectancy differences, but this does not blind allocation. To mitigate bias, we use centralized randomization, standardized instructions, and prespecified analyses; where feasible, data analysts will be masked to group labels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-LMST Intervention (Experimental): Participants use a Meta Quest 3 headset to complete an interactive virtual reality simulation of a rural clinic visit with a Veteran avatar at risk for suicide. The simulation incorporates skills in suicide risk identification, firearm and medication safety counseling, and collaborative safety planning.
  Interventions: Behavioral: Virtual Reality Lethal Means Safety Training
- 2D Video Training (Active Comparator): Participants use a VR headset to view a 10-minute 2D video depicting a lethal means safety counseling session with a veteran.
  Interventions: Behavioral: 2D Video Training

INTERVENTIONS:
Behavioral: Virtual Reality Lethal Means Safety Training — An immersive behavioral training program delivered through a Meta Quest 3 virtual reality headset. Participants enter a simulated rural health clinic and interact with a Veteran avatar at risk for suicide. The simulation incorporates realistic dialogue and decision points where providers practice skills in suicide risk identification, lethal means safety counseling (firearm and medication storage), and collaborative safety planning. The VR format allows repeated practice in a safe environment and provides a more engaging and realistic training experience than traditional methods.
  Arms: VR-LMST Intervention
Behavioral: 2D Video Training — A 10-minute video delivered through a VR headset that depicts a healthcare provider conducting lethal means safety counseling with a Veteran. This is a non-interactive training used as an active comparator.
  Arms: 2D Video Training

SUMMARY:
The goal of this randomized clinical trial is to determine whether a virtual reality (VR) training program can help healthcare providers improve their skills in discussing suicide prevention and safe storage of firearms and medications with Veterans. The study will test whether VR training increases providers' self-efficacy, confidence, and comfort in conducting lethal means safety counseling, and whether it improves their intention to use these counseling practices in their clinical work. Researchers will compare healthcare providers who complete the VR training to those who complete a 2D video training to determine whether the VR approach is more effective. Participants will complete online surveys before and after the training and again three months later. They will be randomly assigned to one of two groups: VR training group: Participants use a VR headset to interact with a virtual Veteran patient in a simulated rural clinic and practice suicide prevention counseling skills; Video training group: Participants use the same headset to watch a ~10-minute 2D video depicting the lethal means safety counseling session. After the training, participants will also provide feedback about their experience, including how realistic and useful they found the training.

DETAILED DESCRIPTION:
This study will test whether a virtual reality (VR) training program can improve healthcare providers' ability to talk with Veterans about suicide prevention and safe storage of firearms and medications. Rural Veterans have suicide rates much higher than the national average, and providers in rural areas often do not receive enough training in suicide risk identification or lethal means safety counseling.

This project builds on our prior Veteran Suicide Assessment in Virtual Reality (VET-SAVR) study, which showed that VR can be a feasible and acceptable way to deliver suicide prevention training. In the current study, called the Virtual Reality Lethal Means Safety Training (VR-LMST) project, we will compare an immersive VR training simulation to a 2D video training.

Study Aims

Aim 1: Develop a VR training simulation focused on suicide prevention counseling with rural Veterans.

Aim 2: Test whether VR-LMST improves provider confidence (primary), and comfortability and intention (secondary) to engage in lethal means safety counseling.

Aim 3: Assess user experience of the VR simulation, including presence, realism, acceptability, feasibility, and tolerability.

Study Design

This is a randomized controlled trial. Participants will be assigned to one of two groups:

VR-LMST group: Participants will use a VR headset (Meta Quest 3) to enter a simulated rural clinic visit with a Veteran avatar who presents with thoughts of suicide. They will practice counseling skills related to safe firearm and medication storage.

2D Video group: Participants will use a VR headset to view a 10-minute video showing a provider having a lethal means safety conversation with a Veteran.

Assessments

Pre-test, post-test, and 3-month follow-up surveys will be completed online.

The Counseling on Access to Lethal Means (CALM) Core Scale (13 items) will measure provider confidence (1-5), comfortability (6-8), and intentions (9-13). An additional two items measure counseling behavior at 3 months (14-15).

The ITC-Sense of Presence Inventory (ITC-SOPI) will measure presence, naturalness, engagement, and negative effects.

Open-ended questions will gather feedback about realism, acceptability, and feasibility.

Demographic and professional background information will also be collected.

Sample Size and Timeline We will recruit 36 participants (18 per group). Power analysis indicates this sample size is sufficient to detect moderate effects with 80% power for the primary outcome.

Phase 1 (completed): Recruited 11 healthcare providers for qualitative interviews; conducted coding and analysis; developed and refined VR and 2D scripts.

Phase 2 (completed): Prototype VR clinic environment developed through iterative meetings with VR developers.

Phase 3 (completed): Pilot playtesting in October 2025 with 5 participants.

Phase 4 (planned): Randomized trial enrollment to begin mid-November 2025.

Phase 5 (planned): 3-month follow-ups to begin January 2026.

Oversight IRB approval was received September 27, 2024, from the University of Texas at Arlington. This study is funded by the American Foundation for Suicide Prevention (AFSP).

Significance This project will test a novel, scalable training method to give allied healthcare providers repeated opportunities to practice suicide prevention counseling in a safe environment. By equipping rural providers with the skills and confidence to have culturally sensitive, Veteran-centered conversations about firearm and medication safety, VR-LMST has the potential to improve clinical practice and reduce suicide risk among rural Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* healthcare providers serving rural Veterans in Texas (e.g., physicians, physician assistants, nurse practitioners, nurses, pharmacists, social workers, healthcare case managers)
* English-speaking
* Able to provide informed consent

Exclusion Criteria:

* Self-reported pregnancy
* History of motor or balance disorders
* Color blindness
* Neurological or cognitive disorders
* Cardiovascular issues that may be worsened by VR use
* Use of cardiac pacemakers, defibrillators, or hearing aids incompatible with VR equipment
* Significant discomfort in virtual reality environments (e.g., severe motion sickness, vertigo)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Confidence in Lethal Means Safety Counseling | Baseline (pre-test), immediately after intervention (post-test), and 3-month follow-up
  Measured by the Counseling on Access to Lethal Means (CALM) Core Scale (Sale et al., 2018) Confidence subscale ("How confident are you that …"). Items are rated on a 4-point scale and summed; higher scores indicate greater confidence (range = 5 - 20).

SECONDARY OUTCOMES:
Comfortability in Lethal Means Safety Counseling | Baseline (pre-test), immediately after intervention (post-test), and 3-month follow-up
  Measured by the Counseling on Access to Lethal Means (CALM) Core Scale (Sale et al., 2018) Comfortability subscale ("How comfortable are you talking about …"). Includes 3 items where 1 = Not Very Comfortable to 4 = Extremely Comfortable. Items are rated on a 4-point scale and summed (range = 3 - 12). Higher scores indicating greater comfort initiating suicide or means-restriction discussions.
Counseling Intentions | Baseline (pre-test), immediately after intervention (post-test), and 3-month follow-up
  Measured by the Counseling on Access to Lethal Means (CALM) Core Scale (Sale et al., 2018) Counseling Intentions subscale ("If you recognize warning signs of suicide in an individual, how likely are you to…"). Includes 5 items where 1 = Not Very Likely to 4 = Extremely Likely. Items are rated on a 4-point scale and summed (range = 5-20). Higher scores indicate stronger intentions to engage in suicide-prevention and lethal-means safety counseling behaviors.
Spatial Presence | Immediately after intervention (post-test only)
  Measured by the ITC-Sense of Presence Inventory (Lessiter et al., 2001) Spatial Presence subscale ("During my experience of the displayed environment…"). Includes 19 items (e.g., "I felt as though I was in the same space as the characters and/or objects") rated on a 5-point scale where 1 = Strongly Disagree to 5 = Strongly Agree. Items are averaged to create a mean subscale score (range = 1 - 5). Higher scores indicate a stronger sense of "being there" or physical immersion within the virtual environment.
Engagement | Immediately after intervention (post-test only)
  Measured by the ITC-Sense of Presence Inventory (Lessiter et al., 2001) Engagement subscale ("During my experience of the displayed environment…"). Includes 13 items (e.g., "I felt myself being drawn in") rated on a 5-point scale where 1 = Strongly Disagree to 5 = Strongly Agree. Items are averaged to create a mean subscale score (range = 1 - 5). Higher scores indicate greater emotional and cognitive involvement in the displayed environment.
Ecological Validity / Naturalness | Immediately after intervention (post-test only)
  Measured by the ITC-Sense of Presence Inventory (Lessiter et al., 2001) Ecological Validity / Naturalness subscale ("During my experience of the displayed environment…"). Includes 5 items (e.g., "The scenes depicted could really occur in the real world") rated on a 5-point scale where 1 = Strongly Disagree to 5 = Strongly Agree. Items are averaged to create a mean subscale score (range = 1 - 5). Higher scores indicate greater perceived realism and naturalness of the virtual environment.
Negative Effects (Tolerability) | Immediately after intervention (post-test only)
  Tolerability will be measured by the ITC-Sense of Presence Inventory (Lessiter et al., 2001) Negative Effects subscale ("During my experience of the displayed environment…"). Includes 6 items (e.g., "I felt dizzy," "I felt nauseous") rated on a 5-point scale where 1 = Strongly Disagree to 5 = Strongly Agree. Items are averaged to create a mean subscale score (range = 1 - 5). Higher scores indicate greater discomfort or simulator-related side effects (e.g., dizziness, eyestrain, nausea) and thus, lower tolerability.

OTHER OUTCOMES:
Feasibility of VR Training (Qualitative) | Immediately after intervention (post-test only)
  Feasibility (extent to which the intervention can be successfully used, delivered, or implemented as intended in a real-world setting) will be assessed through open-ended post-training survey questions and short debrief interviews. Participants will provide qualitative feedback on how realistic and useful they perceived the VR simulation (or 2D video) by responding to prompts such as: "What elements could be included to make the VR training more realistic and representative?" and "Please add any comments you'd like to make about your experience with the VR training." Responses will be coded thematically using qualitative analysis software to identify key themes related to feasibility (ease of use, technical functionality, time burden, and perceived fit for training or clinical settings), as well as related dimensions of realism, training value, and applicability to professional practice.
Acceptability (Qualitative) | Immediately after intervention (post-test only)
  Acceptability (extent to which participants find an intervention appropriate, satisfying, and relevant to their professional role or setting) will be measured by open-ended response to "How much do you agree that the VR training was representative of speaking with a veteran experiencing suicide/depression about lethal means safety?" and provide additional open-ended feedback describing their perceptions of training value, satisfaction, and authenticity. Responses will be coded thematically using qualitative analysis software to identify key themes related to acceptability (appropriateness, satisfaction, and perceived usefulness of the training).

CONTACTS AND LOCATIONS:
Overall Officials: Donna L. Schuman, PhD, LCSW, Principal Investigator — University of Texas at Arlington, School of Social Work
Locations (1):
- University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This study collects survey and qualitative data from a small sample of healthcare providers. Because of the limited sample size and potential identifiability of responses, individual participant data (IPD) will not be shared. Aggregate data will be shared in publications and presentations.

REFERENCES:
- [Background] Sale E, Hendricks M, Weil V, Miller C, Perkins S, McCudden S. Counseling on Access to Lethal Means (CALM): An Evaluation of a Suicide Prevention Means Restriction Training Program for Mental Health Providers. Community Ment Health J. 2018 Apr;54(3):293-301. doi: 10.1007/s10597-017-0190-z. Epub 2017 Nov 28. PMID 29185154
- [Background] Hunter AA, DiVietro S, Boyer M, Burnham K, Chenard D, Rogers SC. The practice of lethal means restriction counseling in US emergency departments to reduce suicide risk: a systematic review of the literature. Inj Epidemiol. 2021 Sep 13;8(Suppl 1):54. doi: 10.1186/s40621-021-00347-5. PMID 34517912
- [Background] Hoyt T, Holliday R, Simonetti JA, Monteith LL. Firearm Lethal Means Safety with Military Personnel and Veterans: Overcoming Barriers using a Collaborative Approach. Prof Psychol Res Pr. 2021 Aug;52(4):387-395. doi: 10.1037/pro0000372. Epub 2021 May 20. PMID 34421193
- [Background] Diurba S, Johnson RL, Siry BJ, Knoepke CE, Suresh K, Simpson SA, Azrael D, Ranney ML, Wintemute GJ, Betz ME. Lethal Means Assessment and Counseling in the Emergency Department: Differences by Provider Type and Personal Home Firearms. Suicide Life Threat Behav. 2020 Oct;50(5):1054-1064. doi: 10.1111/sltb.12649. Epub 2020 Jun 29. PMID 32598076
- [Background] Boggs JM, Quintana LM, Powers JD, Hochberg S, Beck A. Frequency of Clinicians' Assessments for Access to Lethal Means in Persons at Risk for Suicide. Arch Suicide Res. 2022 Jan-Mar;26(1):127-136. doi: 10.1080/13811118.2020.1761917. Epub 2020 May 7. PMID 32379012